CLINICAL TRIAL: NCT03720496
Title: Adoptive Immunotherapy for Refractory/Relapsed Non-Hodgkin Lymphoma With CD19-TriCART Cells
Brief Title: Treatment of Refractory/Relapsed Non-Hodgkin Lymphoma With CD19-TriCART Cell Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Timmune Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2018-8
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Non-hodgkin Lymphoma,B Cell
Keywords: CAR-T; TriCAR-T; CD19-TriCAR-T; Non-hodgkin Lymphoma; NHL; CD19-CAR-T
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-TriCAR-T (Experimental): Tri-functional anti-CD19 chimeric antigen receptor transduced autologous T cells will be administered intravenously
  Interventions: Biological: CD19-TriCAR-T

INTERVENTIONS:
Biological: CD19-TriCAR-T — A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by a single infusion of CAR transduced autologous T cells administered intravenously at a target dose of 0.1-1 x 10^6 CAR+ T cells/kg body weight.

SUMMARY:
This is a single arm, open-label, phase Ⅰ study, to determine the safety and efficacy of CD19-TriCAR-T, an autologous tri-functional anti- CD19 chimeric antigen receptor (CAR)-positive T cell therapy, in Refractory/ Relapsed CD19 Positive Non-Hodgkin Lymphoma (NHL).

DETAILED DESCRIPTION:
The tri-functional anti-CD19 chimeric antigen receptor contains an anti-CD19 scFv, a PD-L1 blocker, and a cytokine complex, enabling the CD19-TriCAR-T to simultaneously targeting the CD19 positive NHL cells，blocking the inhibitory PD-L1 signal and stimulating T/NK cell activation and expansion.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must personally sign and date the consent form before initiating any study specific procedures or activities;
2. All subjects must be able to comply with all the scheduled procedures in the study;
3. Histologically or cytologically confirmed CD19 positive non-Hodgkin lymphoma;
4. At least one measurable lesion per revised IWG Response Criteria;
5. Aged 18 to 69 years;
6. Expected survival ≥12 weeks;
7. Eastern cooperative oncology group (ECOG) performance status of ≤2;
8. Systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 4 weeks;
9. All other treatment induced adverse events must have been resolved to

   ≤grade 1;
10. Laboratory tests must fulfill the following criteria: ANC ≥ 1000/uL, HGB >70g/L, Platelet count ≥ 50,000/uL, Creatinine clearance ≤1.5 ULN, Serum ALT/AST ≤2.5 ULN, Total bilirubin ≤1.5 ULN (except in subjects with Gilbert's syndrome);

Exclusion Criteria:

1. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management. Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment;
2. Patients with symptomatic central nervous system metastasis, intracranial metastasis, and cancer cells found in cerebrospinal fluid are not recommended to participate in this study. Symptom free or post-treatment stable disease or disappearance of lesions should not be excluded. The specific selection is ultimately determined by the investigator;
3. Lactating women;
4. Active infection with hepatitis B (HBsAG positive) or hepatitis C virus (anti-HCV positive);
5. Known history of infection with HIV;
6. Subjects need systematic usage of corticosteroid;
7. Subjects need systematic usage of immunosuppressive drug;
8. Planed operation, history of other related disease, or any other related laboratory tests restrict patients for the study;
9. Other reasons the investigator think the patient may not be suitable for the study.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
safety （Incidence of treatment-related adverse events as assessed by CTCAE v4.03） | 24 months
  Incidence of treatment-related adverse events as assessed by CTCAE v4.03

SECONDARY OUTCOMES:
Complete response rate[CR] (Complete response rate per the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma) | 24 months
  Complete response rate per the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma
Partial response rate [PR] （Partial response rate per the revised International Working Group (IWG) Response Criteria） | 24 months
  Partial response rate per the revised International Working Group (IWG) Response Criteria
Duration of Response （The time from response to relapse or progression） | 24 months
  The time from response to relapse or progression
Progression Free Survival （The time from the first day of treatment to the date on which disease progresses） | 24 months
  The time from the first day of treatment to the date on which disease progresses
Overall Survival （The number of patient alive, with or without signs of cancer） | 24 months
  The number of patient alive, with or without signs of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Lin, Principal Investigator — The Second Affiliated Hospital of Hainan Medical University
Locations (1):
- The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Locke FL, Neelapu SS, Bartlett NL, Siddiqi T, Chavez JC, Hosing CM, Ghobadi A, Budde LE, Bot A, Rossi JM, Jiang Y, Xue AX, Elias M, Aycock J, Wiezorek J, Go WY. Phase 1 Results of ZUMA-1: A Multicenter Study of KTE-C19 Anti-CD19 CAR T Cell Therapy in Refractory Aggressive Lymphoma. Mol Ther. 2017 Jan 4;25(1):285-295. doi: 10.1016/j.ymthe.2016.10.020. Epub 2017 Jan 4. PMID 28129122
- [Background] Neelapu SS, Tummala S, Kebriaei P, Wierda W, Gutierrez C, Locke FL, Komanduri KV, Lin Y, Jain N, Daver N, Westin J, Gulbis AM, Loghin ME, de Groot JF, Adkins S, Davis SE, Rezvani K, Hwu P, Shpall EJ. Chimeric antigen receptor T-cell therapy - assessment and management of toxicities. Nat Rev Clin Oncol. 2018 Jan;15(1):47-62. doi: 10.1038/nrclinonc.2017.148. Epub 2017 Sep 19. PMID 28925994
- [Background] Kalos M, Levine BL, Porter DL, Katz S, Grupp SA, Bagg A, June CH. T cells with chimeric antigen receptors have potent antitumor effects and can establish memory in patients with advanced leukemia. Sci Transl Med. 2011 Aug 10;3(95):95ra73. doi: 10.1126/scitranslmed.3002842. PMID 21832238